CLINICAL TRIAL: NCT05220319
Title: CORTERAS STUDY: The Effect of Corticosteroids on Early Recovery After Major Surgery in Elderly Patients
Acronym: CORTERAS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ziekenhuis Oost-Limburg (Other)
Responsible Party: Principal Investigator, Steven Thiessen, Principal Investigator, Ziekenhuis Oost-Limburg
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Z-2021070
Record Dates: First submitted 2022-01-31; First posted 2022-02-02 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Inflammatory Response; Weakness, Muscle
MeSH Terms: conditions — Muscle Weakness | interventions — Methylprednisolone; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): 100 ml of NaCl 0,9%, not containing corticosteroids, given at induction of anaesthesia, before surgery.
  If a patient will receive cardiopulmonary bypass (CPB) during his operation, a repeat dose of 100 ml of NaCl 0,9% will be administered at the beginning of CPB.
  Interventions: Drug: NaCl 0.9%
- Methylprednisolone (Active Comparator): 250 mg of methylprednisolone made up with 100 ml NaCl 0,9%, given at the induction of anaesthesia, before surgery.
  If a patient will receive cardiopulmonary bypass (CPB) during his operation, a repeat dose of 250 mg methylprednisolone will be administered at the beginning of CPB.
  Interventions: Drug: Methylprednisolone

INTERVENTIONS:
Drug: Methylprednisolone — 250 mg Methylprednisolone made up with 100 ml NaCl0,9% as an IV injection at the induction of anaesthesia but before surgery. If CPB is required an additional dose in 100 ml will be given.
  Arms: Methylprednisolone
Drug: NaCl 0.9% — 100 ml NaCl0,9% as an IV injection at the induction of anaesthesia but before surgery. If CPB is required an additional 100ml will be given.
  Arms: Placebo

SUMMARY:
Major surgery induces a systemic inflammatory response, which can influence the post-operative morbidity, such as coagulation disorders and post-operative muscle weakness, hampering early recovery after surgery.

Single administration of high dose corticosteroids is known to reduce this inflammatory response and could possibly improve the post-operative outcome.

The CORTERAS study will evaluate the effect of administration of corticosteroids, as compared to no corticosteroids, on postoperative muscle weakness and quality of recovery after surgery in elderly patients.

DETAILED DESCRIPTION:
The number of elderly patients undergoing surgery is expected to increase in the coming years, due to the increase in life expectancy in the developing world. Compared to younger surgical patients, the older patients are at greater risk of mortality and morbidity after surgery.

Post-operative fatigue is an important complication after surgery. Not only is it reported by patients as one of the most distressing symptoms, it is also thought to be a significant contributor to delayed recovery after surgery. From a pathophysiological point of view, muscle weakness could be a major contributor to this post-operative fatigue.

Recent studies showed a profound reduction in muscle strength after surgery in elderly patients, which lasted for more than 3 months after surgery. This decrease in muscle strength might be induced by an excessive inflammatory response to surgery.

Glucocorticosteroids are capable of tampering an excessive inflammatory response to surgery and could improve the quality of recovery after surgery. However, a possible effect on post-operative muscle weakness hasn't been specifically investigated.

Therefore, the main objective of this prospective clinical trial is to evaluate the effect of corticosteroids on early post-operative outcome, focusing on muscle weakness, in elderly patients (≥60 years) undergoing surgery.

ELIGIBILITY:
Inclusion Criteria:

* Aged 60 years or older.
* Scheduled for one of the predefined surgical procedures:

  * off-pump coronary bypass surgery
  * on-pump coronary bypass surgery
  * aortic and mitral valve replacement
  * laparoscopic hemicolectomies
  * thoracoscopic lung resections
  * femoral popliteal and tibial bypass surgery and femoral profundoplasty
  * laparoscopic radical prostatectomies

Exclusion Criteria:

* Lack of informed consent or inability to give informed consent.
* Severe postoperative nausea & vomiting (PONV), needing corticosteroids as PONV prophylaxis.
* Urgent, not elective surgery
* Hypersensitivity or known allergic reactions to methylprednisolone
* Preoperative systemic use of steroids:

  * Including, but not limited to, the use of corticosteroids > 4 weeks before surgery of at least 4 mg methylprednisolone equivalents.
  * Excluding inhalational and topical steroids
* Preexisting muscle disease o Including, but not limited to: Steinert's disease, amyotrophic lateral sclerosis (ALS), Duchenne dystrophy, amputation of dominant arm or hand.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 751 (Actual)
Dates: Start 2022-02-16 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-10-28 (Actual)

PRIMARY OUTCOMES:
Post operative muscle weakness | Pre-operative and Post operative day 1
  decrease in muscle strength post-operatively, assessed by comparing the handgrip strength of the dominant hand, measured by the JAMAR dynamometer, on day 1 following surgery as compared to the preoperative value

SECONDARY OUTCOMES:
Post operative muscle weakness | Pre-operative and Post operative day 1, 3 and 5
  Decrease in muscle strength post-operatively, assessed by comparing the handgrip strength of the dominant hand, measured by the JAMAR dynamometer, on day 3 and 5 following surgery as compared to the preoperative value, if still in the hospital.
Maximum inspiratory pressure as measure of respiratory muscle function | Pre-operative and Post operative day 1, 3 and 5
  Maximum inspiratory pressure on day 1, 3 and 5, as compared to pre-operative value, if still in the hospital.
Post operative fatigue | Pre-operative and Post operative day 1, 3, 5 and 28
  Assessed by the Chalder fatigue Questionnaire - 11 items, scores min 0 - max 33, higher score means worse outcome: post-operative day 1, 3, 5 and 28, as compared to preoperatively
Quality of recovery (QOR) | Post operative day 1, 3 and 5
  Assessed by the QOR-15 scale, scores min 0 - max 150, higher score means worse outcome, assessed on day 1, 3 and 5 as compared to preoperatively
Functioning at day 28 | Pre-operative and Post operative day 28
  EuroQol five dimensions of health (EQ5D), score of 1-5 on each health dimension, higher score means worse outcome + visual analogue scale from 0-100 questionning todays health, lower score means worse outcome. EQ5D is assessed on day 28, as compared to pre-operatively values
Coagulation disorder | postoperatively first 24 hours
  biochemical markers of coagulation postoperatively as compared to preoperatively
Sleeping pattern | 10 consecutive nights, starting 3 days before surgery
  Assessed by the Consensus Sleep Diary (CSD) in a subset of study population
Sleep quality | 3 days before and 10 days after surgery
  Assessed by the Pittsburgh Sleep Quality Index (PSQI) in a subet of study population, score range between 0 and 21, higher scores indicate worse sleep quality
Sleep chronotype | 3 days before surgery
  Assessed by the Munich Chronotype Questionnaire (MCTQ) is a subset of study population
Sleeping EEG pattern | first postoperative night
  Assessed by EEG recording in a subset of study population

CONTACTS AND LOCATIONS:
Locations (1):
- Ziekenhuis Oost-Limburg, Genk, Belgium

IPD SHARING:
Plan to Share IPD: No